CLINICAL TRIAL: NCT04958486
Title: Combination Intraventricular Chemotherapy Pilot Study: 5-Azacytidine (5-AZA) and Trastuzumab Infusions Into the Fourth Ventricle or Resection Cavity in Children and Adults with Recurrent or Residual Posterior Fossa Ependymoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David Ilan Sandberg, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0231
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Fossa Ependymoma
Keywords: 5-Azacytidine; Trastuzumab
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: 5-Azacytidine and trastuzumab infusion

INTERVENTIONS:
Drug: 5-Azacytidine and trastuzumab infusion — Patients will receive once weekly 10 mg intraventricular 5-Azacytidine infusions for six consecutive weeks followed by observation in the infusion suite for a minimum of 30 minutes and once weekly 21 mg intraventricular trastuzumab infusions for six consecutive weeks followed by observation for a minimum of 2 hour after each infusion for the first 2 infusions. During this monitoring period, temperature, blood pressure, heart rate, and oxygen saturation will be measured. Patients will also have a neurological examination performed to observe for neurological changes. All patients will undergo an MRI of the brain and total spine with and without gadolinium within 7 days after the final 5-AZA and trastuzumab infusion to determine treatment response and to assess for any signal changes in the brain or spine caused by the infusions and they will have a 30 day and a 90 day follow-up assessment by telephone or in person for assessment of outcome measures and safety

SUMMARY:
The purpose of this study is to establish the safety and tolerability of simultaneous infusions of 5-Azacytidine and trastuzumab into the fourth ventricle of the brain or resection cavity in patients with recurrent posterior fossa ependymoma and to assess the antitumor activity of simultaneous infusions of 5-Azacytidine and trastuzumab into the fourth ventricle of the brain or resection cavity in patients based upon imaging studies and lumbar cerebrospinal fluid (CSF) cytology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified ependymoma, with recurrence or progression anywhere in the brain and/or spine. Patients are also eligible if they have refractory disease, which will be defined as residual tumor which has not been completely cleared despite prior treatments. To be eligible, patients' disease must have originated in the posterior fossa of the brain
* Patient must have either measurable or evaluable tumor as assessed by MRI of the brain and total spine
* An implanted catheter in the fourth ventricle or posterior fossa tumor cavity attached to a ventricular access device or agreement to have one placed.
* A minimum of 4 weeks between any prior radiation treatments or bevacizumab infusions and first infusion of 5-azacytidine or trastuzumab infusions. A minimum of 2 weeks between last dose of any other systemic chemotherapy and first infusion of 5-azacytidine or Trastuzumab into fourth ventricle
* Life expectancy of at least 12 weeks in the opinion of the principal investigator
* Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age
* Existing neurological deficits must have been stable for a minimum of 1 week prior to study enrollment
* Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy
* Adequate bone marrow function defined by peripheral absolute neutrophil count (ANC) ≥ 500/µL, platelet count ≥ 50,000/µL (transfusion independent), and hemoglobin ≥ 9.0 gm/dL (may receive red blood cell (RBC) transfusions)
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.
* Patient with abnormal cardiac function (Shortening fraction less than 28% on echocardiogram) will need cardiology clearance prior to enrollment
* Normal renal and liver function on basic metabolic panel. Any patients with abnormal blood urea nitrogen (BUN), creatinine, alanine aminotransferase(AST) or aspartate aminotransferase (ALT) levels will need nephrology and/or gastroenterology clearance prior to enrollment

Exclusion Criteria:

* Enrolled in another treatment protocol
* Patients with disease that is completely resectable
* Has received another investigational or chemotherapy agent within 2 weeks or radiation therapy within 4 weeks prior to 5-azacytidine or trastuzumab infusion into the fourth ventricle
* Patients with any cardiac issues who are not cleared by cardiology for participation in the study
* Evidence of untreated infection
* Pregnant or lactating women

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Number of patients with new neurological deficits | 7 days after treatment
  A new neurological deficit will be defined as new cranial neuropathy, change in level of consciousness, motor weakness, gait change or cerebellar finding (ataxia, dysmetria, dysdiadochokinesis) that is attributed by treating physicians to infusions. New neurological deficits graded as Grade 3 or higher after infusions will be defined as serious adverse events (SAE's)

SECONDARY OUTCOMES:
Change in disease progression as assessed by magnetic resonance imaging (MRI) | Baseline(before start of treatment),end of treatment (7 days after treatment)
Change in disease progression as assessed by lumbar CSF cytology | Baseline(before start of treatment),end of treatment (7 days after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: David I Sandberg, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No